CLINICAL TRIAL: NCT05896475
Title: Why do Asymptomatic Rotator Cuff Tears Become Painful? Effect of Biomechanical, Psychosocial and Painrelated Factors.
Brief Title: Risk Factors for Asymptomatic Rotator Cuff Tears to Become Symptomatic.
Status: Recruiting | Type: Observational
Sponsor: University Ghent (Other)
Responsible Party: Sponsor
Other Study IDs: ONZ-2023-0062; BOF22/DOC/005 (Other Grant/Funding Number: Bijzonder Onderzoeksfonds (BOF))
Record Dates: First submitted 2023-05-31; First posted 2023-06-09 (Actual); Last update posted 2024-07-15 (Actual); Status verified 2024-07

CONDITIONS: Rotator Cuff Tears
Keywords: Asymptomatic rotator cuff tears; Symptom registration; Observational study
MeSH Terms: conditions — Rotator Cuff Injuries

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 2 Years
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
In this prospective study, subjects older than 55 years with a degenerative asymptomatic rotator cuff tears will be followed for a period of 2 years. After testing, a symptom registration form will be filled in every 3 months. The test moment consists of pain measurements (pain pressure thresholds and conditioned pain modulation), biomechanical measurements (strength (including hand grip strength), range of motion, ultrasound (while measuring electromyographic activity) and shear wave elastography) and psychosocial measurements (psychosocial questionnaires).

DETAILED DESCRIPTION:
In this prospective study, the aim is to determine the risk factors for developing a symptomatic rotator cuff (RC) tear. It is still unknown why some patients with a RC tear develop complaints and others do not. Better understanding of the etiological factors that underlie RC pathology will increase the efficacy of early clinical intervention. A prospective study with a minimum of 2 year follow-up will be conducted. Biomechanical, psychosocial and painrelated factors will be screened as possible risk factors. We hypothesize that negative psychosocial factors and biomechanical impairments will be risk factors for an asymptomatic tear to become symptomatic over time.

ELIGIBILITY:
Inclusion Criteria:

* 55+ years old
* male or female
* asymptomatic rotator cuff tear diagnosed with ultrasound by a medical doctor
* mean visual analogue score (VAS) of < 3 during daily life activities
* no shoulder complaints having a significant influence on daily life activities

Exclusion Criteria:

* recent shoulder trauma
* massive rotator cuff tears
* small partial thickness tears
* neck complaints
* history of shoulder surgery
* history of proximal upper arm fracture
* frozen shoulder
* inflammatory arthritis
* peripheral or central disorders
* cognitive disorders

Ages: 55 Years to 100 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: 55+ years old subjects with an asymptomatic rotator cuff tear
Sampling Method: Probability Sample
Enrollment: 207 (Estimated)
Dates: Start 2023-06-02 (Actual); Primary Completion 2025-06 (Estimated); Study Completion 2026-10 (Estimated)

PRIMARY OUTCOMES:
Pressure Pain Thresholds (PPT) | Baseline - 2 year if remaining asymptomatic or at moment of becoming symptomatic
  PPTs will be measured on three local locations around the shoulder (supraspinatus, infraspinatus and posterior deltoid). Additionally, two more distal PPTs will be measured (erector spinae and triceps surae).
Acromiohumeral distance (AHD) | Baseline - 2 year if remaining asymptomatic or at moment of becoming symptomatic
  The AHD is the shortest linear distance between the inferior edge of the acromion and the superior edge of the humeral head. This will be measured during rest and during muscle activity.

SECONDARY OUTCOMES:
Clinical tests - mobility | Baseline - 2 year if remaining asymptomatic or at moment of becoming symptomatic
  Passive and active scaption - passive external rotation in supine position with arm in 90° abduction - passive internal rotation in supine position with arm in 90° abduction.
Clinical test - strength | Baseline - 2 year if remaining asymptomatic or at moment of becoming symptomatic
  45° scapular elevation - external rotation - internal rotation - hand grip strength
Conditioned Pain Modulation (CPM) | Baseline - 2 year if remaining asymptomatic or at moment of becoming symptomatic
  The conditioning stimulus will comprise of immersion of the foot until the proximal ankle (level of the malleoli) in a hot circulating water bath of 45.5°C during 1 minute. The test stimulus will comprise of pressure pain threshold (PPT) assessments (as described above) before and after completion of the conditioning stimulus.
Central Sensitization Inventory (CSI) | Baseline - 2 year if remaining asymptomatic or at moment of becoming symptomatic
  The CSI measures the participant's Central Sensitization Syndrome related symptoms. The higher the score, the more signs of central sensitization are present.
Tampa Scale for Kinesiophobia (TSK) | Baseline - 2 year if remaining asymptomatic or at moment of becoming symptomatic
  The TSK evaluates the general pain related fear of movement. The higher the score, the higher the pain related fear.
Short Form-36 (SF-36) | Baseline - 2 year if remaining asymptomatic or at moment of becoming symptomatic
  The SF-36 evaluates the general health and well-being or quality of life. Contains a physical and mental component score. A higher score expresses a better health condition.
Shoulder Pain and Disability Index (SPADI) | Baseline - 2 year if remaining asymptomatic or at moment of becoming symptomatic
  The SPADI evaluates the pain and restrictions in activities. The higher the score, the worse the symptoms.
Depression, anxiety and stress scale (DASS-21) | Baseline - 2 year if remaining asymptomatic or at moment of becoming symptomatic
  DASS-21 evaluates the depression (7 items); anxiety (7 items) and stress (7 items). The score will be multiplied by 2 to have a comparable score with the DASS-42.
International Physical Activity Questionnaire (IPAQ) | Baseline - 2 year if remaining asymptomatic or at moment of becoming symptomatic
  The IPAQ will be used to evaluate the physical activity level of the participants. This questionnaire contains 31 questions in 5 domains: 1) physical activity during work; 2) physical activity concerning transport; 3) physical activity by doing household chores; 4) physical activity concerning sport activities; 5) sitting time.
Insomnia Severity Index (ISI) | Baseline - 2 year if remaining asymptomatic or at moment of becoming symptomatic
  Seven questions to ask for sleep problems.
General Self-Efficacy Scale (GSES) | Baseline - 2 year if remaining asymptomatic or at moment of becoming symptomatic
  The GSES measures (10 statements) how a person deals with stressors/difficult situations in life. The scale is about a person's self-confidence that his or her actions are responsible for successful outcomes or, in other words, that one has control over challenging demands imposed by the environment.
Electromyographic activity (EMG) | Baseline - 2 year if remaining asymptomatic or at moment of becoming symptomatic
  Electromyographic activity will be measured during AHD measurement in rest and during activity. The amplitude of the EMG activity from the three parts of the deltoid (anterior, middle and posterior part) will be obtained. The unit is volt. EMG activity will be expressed as percentage of the MVIC (maximal voluntary isometric contraction).
Shear Wave Elastography (SWE) | Baseline - 2 year if remaining asymptomatic or at moment of becoming symptomatic
  This is a non-invasive and real time assessment of tissue mechanical properties that measures the elasticity of the muscles/tendons. The higher the shear modulus/young modulus/shear wave speed, the higher the stiffness. SWE assessment will be done for the followings muscles: supraspinatus, infraspinatus, anterior and posterior deltoid.
Supraspinatus muscle thickness | Baseline - 2 year if remaining asymptomatic or at moment of becoming symptomatic
  The supraspinatus muscle thickness will be measured on two locations: 1) midpoint of the line cranial to the spina scapula; 2) 2 cm medial to the midpoint of the line cranial to the spina scapulae. One longitudinal and one transverse measurement at each of the scanning sites will be performed. This will be measured in mm.
Humeral glenoid distance (HGD) | Baseline - 2 year if remaining asymptomatic or at moment of becoming symptomatic
  The HGD is the distance between the most posterior point of the humeral head and the posterior glenoid. This will be measured in mm.

CONTACTS AND LOCATIONS:
Overall Officials: Alexander Van Tongel, Prof. dr., Principal Investigator — Orthopaedics and Traumatology Ghent University Hospital
Locations (1):
- Department of rehabilitation sciences, Ghent, Oost-Vlaanderen, Belgium